CLINICAL TRIAL: NCT04125654
Title: Clinical Metagenomic Next-Generation Sequencing for Diagnosis of Ascites Infection in End-stage Liver Diseases
Brief Title: Metagenomic Next-Generation Sequencing for Diagnosis of Ascites Infection in End-stage Liver Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); The First Hospital of Jilin University (Other); Beijing Ditan Hospital (Other); Shanghai Public Health Clinical Center (Other Government); Taihe Hospital (Other); Xiangya Hospital of Central South University (Other); Southwest Hospital, China (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The Second Hospital of Shandong University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 010
Record Dates: First submitted 2019-10-07; First posted 2019-10-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Ascites Infection
Keywords: Ascites infection; ascites; mNGS
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with ascites enrolled for mNGS testing (Experimental): Patients with ascites will be enrolled in this study in order to analyze the clinical utility of mNGS for pathogen detection. There is no control group for this study (Investigators will identify historical controls by retrospective clinical documents).
  Interventions: Device: mNGS for pathogen detection

INTERVENTIONS:
Device: mNGS for pathogen detection — This assay is a metagenomic test undertaken by BGI Genomics Co., Ltd. for comprehensive detection of viruses, bacteria, fungi, and parasites in clinical samples.
  Other Names: metagenomic next-generation sequencing testing

SUMMARY:
Ascites is the most common complication of cirrhosis, and its development is associated with substantially increased mortality. Ascites infection including spontaneous bacterial peritonitis (SBP), bacterascites and fungal infections. SBP is one of the most feared complications of ascites. The EASL guidelines recommend that diagnostic criteria of SBP is defined on the ascitic fluid polymorphonuclear leucocytes (PMN) count ≥250 cell/μl, with or without ascites fluid positive culture. However, in clinical practice. Up to 30% of hospitalized patients are considered as suspicious SBP, and treated as SBP without a laboratory-confirmed cause of infection. and is present in 10-30% of all hospitalized patients with ascites. Besides, fungal infection in ascites was aslo related to high mortality in cirrhosis patients.

Thus, to diagnose ascites infection promptly is the key step to prevent the complication. Since, the sensitivity of bacterial culture is limited even if ascites is directly injected into blood culture bottles at the besides. New method to identified the pathogen is needed.

Here, we aim to use metagenomic next-generation sequencing(mNGS) to provide the first-ever demonstration of precision medicine for the diagnosis of ascites infection in hospitalized patients, with immediate impact on clinical care and patients outcomes. The method of mNGS is undertaken by BGI Genomics Company which is a licensed clinical diagnostic laboratory in China. In this multicenter and prospective clinical study, we are planning to detect ascites sample by mNGS and compare the performance of mNGS and routine microbiological testing. Ultimately, we aim to improve the diagnosis of ascites infection and improve patients' outcomes.

DETAILED DESCRIPTION:
The study is divided into 2 parts:

Firstly, the study will test 3 types of sample by means of mNGS, including ascites fluid, peritoneal dialysis fluid and postoperative drainage fluid and evaluate the sensitivity and specificity of NGS.

Secondly, the clinical validation of mNGS will be performed in multicenters for ascites infection in cirrhosis patients. Furthermore, the study will collect the paired plasma sample for NGS testing at the same time to evaluate the protential sources of microorganisms in ascites.The aim of the study is to observe the performance of mNGS in ascites infection diagosis and the protential clinical effect in cirrhsis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization cirrhotic patients;
2. Age >18 years old;
3. Paitents with ascites at hospital admission.

Exclusion Criteria:

1. Pregnant women;
2. Hepatic tumor or extrahepatic related cancer;
3. Identified secondary peritonitis;
4. Ascites not related to portal hypertension;
5. Not provide written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical mNGS assay performance (mNGS positive number and the pathogenics species) | within 1 month of patient enrollment in study
  mNGS positive number and the pathogenics species in ascites
Classification of ascites infection based on mNGS result. | within 1 month of patient enrollment in study.
  Proportion of spontaneous bacterial peritonitis, bacterascites, neutrocytic ascites and sterile ascites based on mNGS result.

SECONDARY OUTCOMES:
The proportion of acute kindey injury. | within 1 month of patient enrollment in study.
  The proportion of acute kindey injury between ascites NGS positive and negative groups.
90-day mortality | within 90 days of patient enrollment in study
The proportion of new-onset spontaneous bacterial peritonitis. | within 1 month of patient enrollment in study.

CONTACTS AND LOCATIONS:
Overall Officials: Aishan Su, Study Director — Nanfang Hospital Guangzhou, Guangdong, China, 510515
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China